#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for A Phase I, Open-Label, Single-Dose, Two-Part Study to Assess the Pharmacokinetics of Gepotidacin (GSK2140944) in Male and Female Adult Participants with Varying Degrees of Hepatic Impairment and in Matched Control Participants with Normal Hepatic Function |
| <b>Compound Number</b> | : | GSK2140944 |
| <b>Effective Date</b> | : | 29-JUN-2018 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol BTZ117352.
- This RAP is intended to describe the safety, tolerability, and pharmacokinetic (PK) analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) and Interim Analysis (IA) deliverable.

#### **RAP Author(s):**

| PPD | 20 HIN 2010 |
|---|---|
| Biostatistician II (Biostatistics, Early Development Services, PPD) | 29-JUN-2018 |
| PPD | 29-JUN-2018 |
| Pharmacokineticist (Biostatistics, PPD) | 29-JUN-2018 |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Principal Statistician (Infectious Disease,<br>Clinical Statistics) | 29-JUN-2018 | Email |
| Principal Programmer/ Analyst (Infectious Disease, Clinical Statistics) | 27-JUN-2018 | Email |
| SM Executive Medical Director (Infectious Disease, RD ID) | 27-JUN-2018 | Email |
| Clinical Development Director (Infectious Disease, RD PCPS Therapy Area Delivery ID) | 27-JUN-2018 | Email |
| Manager (Clinical Data Management) | 29-JUN-2018 | Email |
| PPD Director (Clinical Pharmacology) | 27-JUN-2018 | Email |
| Director (GCSP Medical SERM US) | 27-JUN-2018 | Email |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| PPD | 27-JUN-2018 | Email |
| Director (Infectious Disease, Clinical Statistics) | | - |
| PPD | | |
| Programming Manager (Infectious Disease,<br>Clinical Programming) | 28-JUN-2018 | Email |

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | INTRO | DUCTIO | DN | | 5 |
| 2. | SLIMM | IARY OF | KEY PROT | TOCOL INFORMATION | 5 |
| ۷. | 2.1. | | | tocol Defined Statistical Analysis Plan | |
| | 2.2. | | | and Endpoint(s) | |
| | 2.3. | | | | |
| | 2.4. | | | | |
| 3. | PLANI | NED AN | ALYSES | | 10 |
| | 3.1. | | | | |
| | 3.2. | | | | |
| 4. | ANALY | /SIS PO | PULATIONS | S | 11 |
| | 4.1. | Protoco | l Deviations | | 11 |
| 5. | | | | DATA ANALYSES AND DATA HANDLING | |
| | | | | 0.1 | |
| | 5.1. | | | Sub-group Display Descriptors | |
| | 5.2.<br>5.3. | | | sns for Data Analyses and Data Handling | 12 |
| | 5.5. | | | is for Data Arialyses and Data Handling | 13 |
| 6. | STUD | Y POPU | I ATION AN | ALYSES | 14 |
| ٥. | 6.1. | | | d Study Population Analyses | |
| 7. | рцирі | MACOK | INIETIC ANIA | ALYSES | 15 |
| 1. | 7.1. | | | kinetic Analyses | |
| | 7.1. | 7.1.1. | | / Variables | |
| | | 7.1.1. | 7.1.1.1. | | |
| | | | 7.1.1.1.<br>7.1.1.2. | Derived Pharmacokinetic Parameters | |
| | | 7.1.2. | | Measure | |
| | | 7.1.3. | • | n of Interest | |
| | | 7.1.4. | | Analyses / Methods | |
| | | | | Statistical Methodology Specification | |
| | 7.2. | Second | | cokinetic Analyses | |
| | | 7.2.1. | | / Variables | |
| | | | 7.2.1.1. | Drug Concentration Measures | |
| | | | 7.2.1.2. | Derived Pharmacokinetic Parameters | |
| | | 7.2.2. | Summary | Measure | |
| | | 7.2.3. | • | n of Interest | |
| | | 7.2.4. | | Analyses / Methods | |
| | | | 7.2.4.1. | Statistical Methodology Specification | |
| | 7.3. | Explora | tory Pharma | acokinetic Analyses | |
| | | 7.3.1. | | / Variables | |
| | | | 7.3.1.1. | Drug Concentration Measures | 19 |
| | | | 7.3.1.2. | Derived Pharmacokinetic Parameters | |
| | | 7.3.2. | Summary | Measure | 20 |
| | | 7.3.3. | Population | n of Interest | |

| | | 7.3.4. | Statistical Analyses / Methods | <mark>20</mark> |
|---|---|---|---|---|
| | | | 7.3.4.1. Statistical Methodology Specification | 20 |
| 8. | SAFF | ΓΥ ΑΝΑΙ ` | YSES | 22 |
| Ο. | 8.1. | | Events Analyses | |
| | 8.2. | | Events of Special Interest Analyses | |
| | 8.3. | | Laboratory Analyses | |
| | 8.4. | | afety Analyses | |
| 9. | REFE | RENCES | | <mark>23</mark> |
| 10. | APPEI | NDICES. | | 24 |
| | 10.1. | | x 1: Schedule of Activities | |
| | | | Protocol Defined Time and Events Table | |
| | | 10.1.2. | Protocol Defined Safety and PK Assessments | |
| | 10.2. | Appendi | x 2: Study Phases and Treatment Emergent Adverse | |
| | | Events | | |
| | | 10.2.1. | | |
| | | | 10.2.1.1. Study Phases for Concomitant Medication | |
| | | 10.2.2. | Treatment Emergent Flag for Adverse Events | |
| | 10.3. | Appendi | x 3: Data Display Standards & Handling Conventions | <mark>29</mark> |
| | | 10.3.1. | 1 3 | |
| | | 10.3.2. | Reporting Standards | <mark>2</mark> 9 |
| | | 10.3.3. | Reporting Standards for Pharmacokinetic | 30 |
| | 10.4. | Appendi | x 4: Derived and Transformed Data | |
| | | 10.4.1. | General | 31 |
| | | 10.4.2. | Study Population | 31 |
| | | 10.4.3. | Safety | 31 |
| | 10.5. | Appendi | x 5: Reporting Standards for Missing Data | 3 <mark>3</mark> |
| | | 10.5.1. | Premature Withdrawals | 3 <mark>3</mark> |
| | | 10.5.2. | Handling of Missing Data | 3 <mark>3</mark> |
| | | | 10.5.2.1. Handling of Missing and Partial Dates | 3 <mark>3</mark> |
| | 10.6. | Appendi | x 6: Values of Potential Clinical Importance | 34 |
| | | 10.6.1. | ECG | 34 |
| | | 10.6.2. | Vital Signs | 34 |
| | 10.7. | Appendi | x 7: Abbreviations & Trade Marks | 3 <mark>5</mark> |
| | | 10.7.1. | Abbreviations | 3 <mark>5</mark> |
| | | 10.7.2. | Trademarks | 36 |
| | 10.8. | Appendi | x 8: List of Data Displays | 37 |
| | | 10.8.1. | Data Display Numbering | |
| | | 10.8.2. | Mock Example Shell Referencing | |
| | | 10.8.3. | Deliverables | 37 |
| | | 10.8.4. | Study Population Tables | |
| | | 10.8.5. | Safety Tables | |
| | | 10.8.6. | Pharmacokinetic Tables | |
| | | 10.8.7. | Pharmacokinetic Figures | |
| | | 10.8.8. | ICH Listings | |
| | | 10.8.9. | Non-ICH Listings | |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol BTZ117352

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan Rationale for Change | |
| Listings for hypersensitivity AEs will be included where an event | Such listings will not be produced regardless of | Tracking of hypersensitivity AEs is not necessary for |
| has occurred | event occurrence | this compound. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare the plasma PK parameters of a 1500 mg oral dose of gepotidacin in normal healthy participants to participants with mild, moderate, and severe hepatic impairment | <ul> <li>Plasma gepotidacin AUC(0-∞) and Cmax, as data<br/>permit.</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>To assess the safety and tolerability of gepotidacin administered as a 1500 mg oral dose in normal healthy participants compared with participants with mild, moderate, and severe hepatic impairment</li> <li>To compare the secondary plasma PK parameters of 1500 mg oral dose of gepotidacin in normal healthy participants with mild, moderate, and severe hepatic impairment</li> <li>To compare the urine PK parameters of a 1500 mg oral dose of gepotidacin in normal healthy participants with participants with</li> </ul> | <ul> <li>12-lead safety ECG readings, change from baseline in vital sign measurements (blood pressure and heart rate), monitoring of AEs, toxicity grading of clinical laboratory test results, and physical examinations</li> <li>Plasma gepotidacin AUC(0-t), Tmax, tlag, CL/F, Vz/F, λz, and t1/2, as data permit</li> <li>Urine gepotidacin PK endpoints: <ul> <li>Primary: Ae total, fe %, and CLr, as data permit</li> <li>Secondary: Ae(t1-t2), AUC(0-12), AUC(0-24), and AUC(0-48), as data permit</li> </ul> </li> </ul> |

| Objectives | Endpoints |
|---|---|
| mild, moderate, and severe hepatic impairment | |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate the saliva PK parameters of a 1500 mg oral dose of gepotidacin in normal healthy participants compared with participants with mild, moderate, and severe hepatic impairment | <ul> <li>Saliva gepotidacin PK endpoints:</li> <li>○ Primary: AUC(0-∞) and Cmax, as data permit</li> <li>○ Secondary: AUC(0-t), Tmax, λz, t1/2, CL/F, Vz/F, and saliva to unbound plasma AUC(0-t) and AUC(0-∞) ratios (RAUC) of gepotidacin, as data permit.</li> </ul> |

#### 2.3. Study Design

#### **Overview of Study Design and Key Features**

# Part 1

Group B: Participants with moderate hepatic impairment

Group D: Participants with normal hepatic function

# PK requirements to continue to Part 2 Observed Mean Values: AUC <48 μg•hr/mL Cmax <14 μg/mL

(Based on emerging data, and/or data that are not expected to exceed these requirements in participants with severe hepatic impairment or may require dose adjustment, participants in Part 2 will be enrolled.)

# Part 2

Group A: Participants with mild hepatic impairment (optional)1

Group C: Participants with severe hepatic impairment<sup>2</sup>

Group E: Participants with normal hepatic function (optional)3

- Based on emergent data from Part 1, participants with mild hepatic impairment (Group A) may not be enrolled in Part 2 if there is not a significant difference between participants with moderate hepatic impairment and participants with normal hepatic function.
- If AUC and/or Cmax are predicted to exceed the threshold, the dose may be adjusted for participants with severe hepatic impairment (Group C). Due to the potential difficulty in identifying eligible participants with severe hepatic impairment, the sponsor may stop the study prior to full enrollment in Part 2 provided that a minimum of 6 evaluable participants with severe hepatic impairment have been enrolled.
- 3. Based on emergent data from Part 1, matching participants with normal hepatic function in Part 2 (Group E) may be enrolled (e.g. if a change in dose is needed or if the demographic data of the mild and/or severe hepatic impairment groups is not well matched to the moderate control data [Group D]).

| Overview of Study Design and Key Features | |
|---|---|
| Design | Phase I, nonrandomized, open-label, parallel-group, multi-center, two- |
| Features | Part study. |
| | <ul> <li>Part 1: Approximately 16 participants, 8 with moderate hepatic impairment (Group B) and 8 matched controls with normal hepatic function (Group D) will receive a single 1500 mg oral dose of gepotidacin. Controls will be matched on gender distribution, age (approximately ± 10 years), and BMI (approximately ± 20%).</li> <li>Part 2: Approximately 8 to 32 participants will receive a single oral dose of gepotidacin. The dose is expected to be 1500 mg, but may be adjusted for participants with severe hepatic impairment if AUC and/or Cmax are predicted to exceed the threshold. Based on emergent data from Part 1, participants with mild hepatic impairment (Group A) may not be enrolled in Part 2 if there is not a significant difference between participants with moderate hepatic impairment and participants with normal hepatic function. Due to the potential difficulty in identifying eligible participants with severe hepatic impairment, the sponsor may stop the study prior to full enrollment in Part 2 provided that a minimum of 6 evaluable participants with severe hepatic </li> </ul> |
| | impairment have been enrolled. Based on emergent data from Part 1, matching participants with normal hepatic function in Part 2 (Group E) may be enrolled (e.g. if a change in dose is needed or if the demographic data of the mild and/or severe hepatic impairment groups is not well matched to the moderate control data [Group D]). |
| Dosing | Participants will receive a single 1500 mg oral dose of gepotidacin delivered as two 750 mg tablets. The dose may be adjusted in Part 2 for participants with severe hepatic impairment if AUC and/or Cmax are predicted to exceed the threshold, based on emergent data from Part 1. |
| Time and Events | See Appendix 1: Schedule of Activities |
| Treatment<br>Assignment | <ul> <li>At Screening, participants will be enrolled to the appropriate groups based on<br/>the classification as defined in the Food and Drug Administration (FDA)<br/>Guidance for Industry, Pharmacokinetics in Patients with Impaired Hepatic<br/>Function: Study Design, Data Analysis, and Impact on Dosing and Labeling<br/>[DHHS, 2003]. Participants with hepatic impairment will be classified using the<br/>Child-Pugh system. For more details, see Section 7.3 of the protocol.</li> </ul> |
| Interim<br>Analysis | <ul> <li>Formal interim analyses of the primary and secondary PK endpoints, will be conducted following completion of Part 1 of the study; with possible progression to Part 2 based on the following criteria: <ul> <li>Participants with mild hepatic impairment may be enrolled in Part 2 if there is a significant difference in pharmacokinetics between participants with moderate hepatic impairment compared with participants with normal hepatic function.</li> <li>Participants with severe hepatic impairment will be enrolled in Part 2 provided that the PK requirements are met (observed mean values in participants with moderate impairment do not exceed the threshold:</li> </ul> </li> </ul> |

| Overview of Study Design and Key Features | |
|---|---|
| | AUC < 48 μg•hr/mL and Cmax < 14 μg/mL). The dose may be adjusted |
| | for participants with severe hepatic impairment if either PK parameter is predicted to exceed the threshold. |
| | <ul> <li>No formal interim analyses of the safety endpoints will be done, but GSK will review the safety data from Part 1 prior to proceeding to Part 2.</li> </ul> |

# 2.4. Statistical Analyses

An estimation approach will be taken to characterize the PK of gepotidacin in subjects with mild, moderate, and severe hepatic impairment compared with matched subjects with normal hepatic function.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

Formal interim analyses of the primary and secondary PK endpoints (as detailed in Section 7.1 and Section 7.2 of this document) will be conducted following completion of Part 1 of the study; with possible progression to Part 2 based on the following criteria:

- Participants with mild hepatic impairment may be enrolled in Part 2 if there is a significant difference in pharmacokinetics between participants with moderate hepatic impairment compared with participants with normal hepatic function.
- Participants with severe hepatic impairment will be enrolled in Part 2 provided that the PK requirements are met (observed mean values in participants with moderate impairment do not exceed the threshold: AUC < 48  $\mu$ g•hr/mL and Cmax < 14  $\mu$ g/mL). The dose may be adjusted for participants with severe hepatic impairment if either PK parameter is predicted to exceed the threshold.

No formal interim analyses of the safety endpoints will be done, but GSK will review the safety data from Part 1 prior to proceeding to Part 2.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Population Definition / Criteria | |
|---|---|---|
| Safety | Consists of all subjects who receive at least 1 dose of study drug and have at least one postdose safety assessment. | <ul><li>Study Population</li><li>Safety</li></ul> |
| PK Population | Consists of all subjects who received at least 1 dose of gepotidacin and have evaluable PK data for gepotidacin. A subject is considered to have evaluable PK data for gepotidacin if the subject has at least 1 measurable post-dose PK concentration value for gepotidacin that was not excluded from the analysis due to a protocol deviation. | PK Concentration |
| PK Parameter | Consist of all subjects in the PK Population, for<br>whom valid and evaluable PK parameters<br>were derived. This population will be used in<br>the assessment and characterization of PK<br>parameters. | <ul><li>PK parameter</li><li>PK statistical analysis</li></ul> |

#### NOTES:

• Please refer to Appendix 8: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarized and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- O Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorized on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the electronic case report form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

#### 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions <sup>[1]</sup> | | | |
|---|---|---|---|---|
| Study | | Hepatic Impairment Group | Data Displays for Reporting | |
| Part | Code | Description | Description | Order <sup>[2]</sup> |
| 1, 2 | D, E <sup>[3]</sup> | Normal Hepatic Function | Normal | 1 |
| 1 | В | Moderate Hepatic Impairment | Moderate | 3 |
| 2 | <b>A</b> <sup>[4]</sup> | Mild Hepatic Impairment (optional) | Mild | 2 |
| 2 | C <sup>[5]</sup> | Severe Hepatic Impairment | Severe | 4 |

#### NOTES:

- 1. Only groups that are present in the data will actually be presented.
- 2. Order represents treatments being presented in TFL, as appropriate.
- 3. Based on emergent data from Part 1, matching participants with normal hepatic function in Part 2 (Group E) may be enrolled (e.g., if a change in dose is needed or if the demographic data of the mild and/or severe hepatic impairment groups is not well matched to the moderate control data [Group D]). If there is no change in dose, then these two groups will be combined for presentation in the outputs.
- 4. Based on emergent data from Part 1, participants with mild hepatic impairment (Group A) may not be enrolled in Part 2 if there is not a significant difference between participants with moderate hepatic impairment and participants with normal hepatic function.
- 5. If AUC and/or Cmax are predicted to exceed the threshold, the dose may be adjusted for participants with severe hepatic impairment (Group C). Due to the potential difficulty in identifying eligible participants with severe hepatic impairment, the sponsor may stop the study prior to full enrollment in Part 2 provided that a minimum of 6 evaluable participants with severe hepatic impairment have been enrolled.

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the last available assessment prior to time of study drug administration, unless noted otherwise.

| Parameter | Study Assess | Baseline Used in<br>Data Display | | |
|---|---|---|---|---|
| | Screening | Screening Day -1 Day 1 (Pre-Dose) | | |
| Safety | | | | |
| Hematology | X | Χ | | Day -1 |
| Clinical Chemistry | X | Χ | | Day -1 |
| 12-Lead ECG | Х | Х | X | Day 1 (Pre-Dose) |
| Vital Signs | X | Х | X | Day 1 (Pre-Dose) |

#### NOTES:

 Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.2 | Appendix 2: Study Phases and Treatment Emergent Adverse Events |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Reporting Standards for Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 8: List of Data Displays.

#### 7. PHARMACOKINETIC ANALYSES

#### 7.1. Primary Pharmacokinetic Analyses

#### 7.1.1. Endpoint / Variables

#### 7.1.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for Pharmacokinetic). Only total gepotidacin plasma PK concentrations will be measured and reported. Therefore, unbound plasma PK concentrations will be derived by multiplying the total plasma PK concentrations by 0.67, to correct for the low plasma protein binding of gepotidacin (33%) observed in previous studies.

#### 7.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-∞) | Area under the concentration-time curve from time 0 (predose) extrapolated to infinite time, calculated as: |
| | $AUC = AUC(0-t) + C(t) / \lambda z$ |
| | where C(t) is the last quantifiable concentration |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data |

#### NOTES:

- Additional parameters may be included as required.
- For the derivation of unbound plasma PK parameters; the total plasma PK parameters AUC(0-∞), and Cmax will be multiplied by 0.67, to correct for the low plasma protein binding of gepotidacin (33%) observed in previous studies.

#### 7.1.2. Summary Measure

Area under concentration-time curve (AUC[ $0-\infty$ ]) and Cmax following single doses of gepotidacin in subjects with normal hepatic function and hepatically impaired subjects.

#### 7.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the PK population for plasma PK concentrations and the PK parameter population for plasma PK parameters and statistical analysis, unless otherwise specified.

#### 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 8: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.1.1 will be summarized using descriptive statistics, graphically presented (where appropriate) and listed

#### 7.1.4.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

#### **Endpoint / Variables**

 Plasma primary pharmacokinetic (PK) endpoints include AUC(0-∞) and Cmax of gepotidacin, as data permit.

#### **Model Specification**

 The plasma In-transformed AUC(0-∞) and Cmax values for gepotidacin in the hepatic impairment groups and the normal hepatic function group will be compared using an analysis of variance (ANOVA).

#### **Model Checking & Diagnostics**

 Model assumptions will be applied, but appropriate adjustments may be made based on the data.

#### **Model Results Presentation**

• Statistical analysis by ANOVA will be presented in tabular format with geometric mean ratios between hepatic impairment groups and normal hepatic function group, and 90% CIs for the ratios of AUC(0-∞) and Cmax for gepotidacin.

# 7.2. Secondary Pharmacokinetic Analyses

#### 7.2.1. Endpoint / Variables

#### 7.2.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for Pharmacokinetic)

#### 7.2.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times.

Plasma pharmacokinetic parameters listed below will be determined from the total plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time 0 (predose) to time of last quantifiable |
| | concentration, to be calculated using the linear trapezoidal rule for each incremental |
| | trapezoid and the log trapezoidal rule for each decremental trapezoid |
| Tmax | Time to first occurrence of Cmax |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| t½ | Terminal half-life will be calculated as: |
| | $t\frac{1}{2} = \ln 2 / \lambda z$ |
| λz | Terminal-phase rate constant |
| CL/F | The apparent oral clearance, calculated as: |
| | CL/F = Dose / AUC(0-∞) |
| Vz/F | The apparent volume of distribution during the terminal phase, calculated as: |
| | $Vz/F = CL / \lambda z$ |

#### NOTES:

- Additional parameters may be included as required.
- For the derivation of unbound plasma PK parameters; the total plasma PK parameters AUC(0-t) will be multiplied by 0.67, and the total plasma PK parameter CL/F will be divided by 0.67, to correct for the low plasma protein binding of gepotidacin (33%) observed in previous studies.

Pharmacokinetic parameters listed will be determined from the urine concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| Ae total | Total unchanged drug (total amount of drug excreted in urine), calculated by adding all the fractions of drug collected over all the allotted time intervals |
| Ae(t1-t2) | Amount of drug excreted in urine in time intervals for predose, 0 to 6, 6 to 12, 12 to 24, 24 to 36, and 36 to 48 hours after dosing for subjects with hepatic impairment; and predose, 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours for subjects with normal hepatic function; calculated by multiplication of the urine concentration for a time interval and the length of this time interval. |
| AUC(0-t) | Area under the urine concentration-time curve over t hours where t = 12, 24, and 48 hours. The AUC(0-t) will be calculated by the linear trapezoidal rule based on the urine concentration data from each collection interval versus the corresponding urine collection interval. |
| Fe% | Percentage of the given dose of drug excreted in urine, calculated as: |
| | fe% = (Ae total/Dose) × 100 |
| CLr | Renal clearance of drug, calculated as: |
| | CLr = Ae total/AUC(0-t) |
| | where AUC(0-t) is the area under the plasma concentration-time curve over all the allotted time intervals of urine collections. |

#### NOTES:

• Additional parameters may be included as required.

#### 7.2.2. Summary Measure

Area under concentration-time curve (AUC[0-48]) and CLr following single doses of gepotidacin in subjects with normal hepatic function and hepatically impaired subjects.

#### 7.2.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the PK population for plasma and urine PK concentrations, and the PK parameter population for plasma and urine PK parameters and statistical analysis, unless otherwise specified.

#### 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 8: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.2.1 will be summarized using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.2.4.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- Plasma secondary PK endpoints include AUC(0-t), Tmax, tlag, CL/F, λz, and t1/2, as data permit.
- Urine primary PK endpoints include AUC(0-48) and CLr of gepotidacin, as data permit. Urine secondary PK endpoints include Ae(t1-t2), AUC(0-12), AUC(0-24), and AUC(0-48) of gepotidacin, as data permit

#### **Model Specification**

- The plasma Tmax will be analyzed non-parametrically using the Mann Whitney U test (Wilcoxon rank sum test). The point estimates and 90% CI for the median differences will be derived for hepatic impairment and healthy participants based on Hodges-Lehmann estimation.
- The urine In-transformed AUC(0-48) and non-transformed CLr values for gepotidacin in the hepatic impairment groups and the normal hepatic function group will be compared using an analysis of variance (ANOVA).

#### **Model Checking & Diagnostics**

 Model assumptions will be applied, but appropriate adjustments may be made based on the data.

#### **Model Results Presentation**

- The point estimates and 90% confidence intervals for the median differences in plasma Tmax will be calculated for the cohort difference (hepatically impaired healthy participants).
- Statistical analysis by ANOVA will be presented in tabular format with geometric mean ratios between hepatic impairment groups and normal hepatic function group, and 90% CIs for the ratios of AUC(0-48) for gepotidacin. For non-transformed CLr for gepotidacin, least squares mean difference between hepatic impairment groups and normal hepatic function group, and 90% CIs for the difference will be presented.

# 7.3. Exploratory Pharmacokinetic Analyses

#### 7.3.1. Endpoint / Variables

#### 7.3.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for Pharmacokinetic)

#### 7.3.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the saliva concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time 0 (predose) to time of last quantifiable concentration, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-∞) | Area under the concentration-time curve from time 0 (predose) extrapolated to infinite time, calculated as: |
| | $AUC(0-\infty) = AUC(0-t) + C(t) / \lambda z$ |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Tmax | Time to first occurrence of Cmax |
| t1/2 | Terminal phase half-life will be calculated as: |
| | $t\frac{1}{2} = \ln 2 / \lambda z$ |
| λz | Terminal-phase rate constant |
| CL/F | The apparent oral clearance, calculated as: |
| | CL/F = Dose / AUC(0-∞) |
| Vz/F | The apparent volume of distribution during the terminal phase, calculated as: $Vz/F = CL / \lambda z$ |
| RAUC(0-t) | The ratio of the AUC(0-t) observed in saliva relative to the unbound AUC(0-t) in plasma, calculated as: |
| | RAUC(0-t) = AUC(0-t) saliva / AUC(0-t) plasma |
| RAUC(0-∞) | The ratio of the AUC( $0-\infty$ ) observed in saliva relative to the unbound AUC( $0-\infty$ ) in plasma, calculated as: |
| | $RAUC(0-\infty) = AUC(0-\infty)$ saliva / $AUC(0-\infty)$ plasma |

#### NOTES:

- Additional parameters may be included as required.
- Since plasma protein binding of gepotidacin is low (33%), only total plasma drug concentrations and total plasma
  PK parameters will be reported for the plasma PK analysis. However, to derive the saliva to unbound plasma
  AUC(0-t) and AUC(0-∞) ratios, a correction factor of 0.67 will be applied to the total plasma AUCs of gepotidacin
  to derive the unbound plasma AUCs.

#### 7.3.2. Summary Measure

Area under concentration-time curve (AUC[ $0-\infty$ ]) and Cmax following single doses of gepotidacin in subjects with normal hepatic function and hepatically impaired subjects.

#### 7.3.3. Population of Interest

The primary pharmacokinetic analyses will be based on the PK population for saliva PK concentrations and the PK parameter population for saliva PK parameters and statistical analysis, unless otherwise specified.

#### 7.3.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 8: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.3.1 will be summarized using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.3.4.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well-defined saliva profiles).

#### **Endpoints**

 Saliva exploratory pharmacokinetic (PK) endpoints include AUC(0-∞), Cmax, and Tmax of gepotidacin, as data permit.

#### **Model Specification**

- The plasma In-transformed AUC(0-∞) and Cmax values for gepotidacin in the hepatic impairment groups and the normal hepatic function group will be compared using an analysis of variance (ANOVA).
- Saliva Tmax will be analyzed non-parametrically using the Mann Whitney U test (Wilcoxon rank sum test). The point estimates and 90% CI for the median differences will be derived for hepatic impairment and healthy participants based on Hodges-Lehmann estimation.

#### **Model Checking & Diagnostics**

 Model assumptions will be applied, but appropriate adjustments may be made based on the data.

#### **Model Results Presentation**

- Statistical analysis by ANOVA will be presented in tabular format with geometric mean ratios between hepatic impairment groups and normal hepatic function group, and 90% CIs for the ratios of AUC(0-∞), Cmax, and AUC(0-48) for gepotidacin.
- Scatter plots of natural In-transformed saliva gepotidacin concentrations versus the natural Intransformed unbound and total plasma gepotidacin concentrations will be plotted and a regression line will be fitted.
- Scatter plots of natural In-transformed saliva gepotidacin PK parameters versus the natural

- In-transformed unbound and total plasma gepotidacin PK parameters will also be performed for the AUC(0-∞), AUC(0-t), Cmax, CL/F, and t1/2.
- The point estimates and 90% confidence intervals for the median differences in Tmax will be calculated for the cohort difference (hepatically impaired healthy participants).

#### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

#### 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 8: List of Data Displays.

#### 8.2. Adverse Events of Special Interest Analyses

Liver monitoring/stopping events and cardiovascular events will be considered AEs of Special Interest (AESIs). AESIs are flagged in the eCRF and details of events are collected on special eCRF pages. The details of the planned displays are provided in Appendix 8: List of Data Displays.

#### 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. Division of Microbiology and Infectious Diseases (DMID) grading for all parameters as specified in the protocol will be assigned programmatically by PPD in the Laboratory Analysis Dataset. DMID grading will be applied for all subjects, regardless of hepatic impairment. The details of the planned displays are in Appendix 8: List of Data Displays.

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 8: List of Data Displays.

#### 9. REFERENCES

Department of Health and Human Services (DHHS), Food and Drug Administration, Center for Drug Evaluation and Research, Center for Biologics Evaluation and Research (US). Guidance for Industry: Pharmacokinetics in Patients with Impaired Hepatic Function: Study Design, Data Analysis, and Impact on Dosing and Labeling. May 2003. [19 screens]. Available from:

https://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm072123.pdf

GlaxoSmithKline Document Number 2017N352027\_00 (Original – 15-FEB-2018): A Phase I, Open-Label, Single-Dose, Two-Part Study to Assess the Pharmacokinetics of Gepotidacin (GSK2140944) in Male and Female Adult Participants with Varying Degrees of Hepatic Impairment and in Matched Control Participants with Normal Hepatic Function (15-FEB-2018)

# 10. APPENDICES

# 10.1. Appendix 1: Schedule of Activities

# 10.1.1. Protocol Defined Time and Events Table

| | Screening<br>(up to | Check-<br>in | Tre | atment Pe<br>(Days) | riod | Follow-up<br>(10 [±5] | |
|---|---|---|---|---|---|---|---|
| Procedure <sup>1</sup> | 30 days<br>prior to<br>Day -1) | -1 | 1 | 1 2 | | days postdose) or Early Termination | Notes |
| Confined to clinic | | Х | Х | X | Х | | Participants will be admitted to the clinic on Day –1 and will be discharged on Day 3. Confinement will be 4 days and 3 overnight stays |
| Informed consent | Х | | | | | | |
| Inclusion and exclusion criteria | Х | Х | | | | | Recheck clinical<br>status before<br>enrollment and/or<br>study drug<br>administration |
| Demographics | Х | | | | | | |
| Complete physical examination including height and weight | Х | | | | | | |
| Abbreviated physical examination | | Х | | | Х | Х | |
| Medical history<br>(includes substance<br>usage and history of<br>hepatic disease) | X | | | | | | Substances: drugs, alcohol, and caffeine. Participants with hepatic impairment should be on a stable regimen of chronic medications 7 days before study drug administration on Day 1 |
| Past and current<br>medical conditions<br>(including hepatic<br>impairment medical<br>history, Child-Pugh<br>score, and Clcr) | X | | | | | | Child-Pugh as defined<br>in the FDA Guidance<br>for Industry:<br>Pharmacokinetics in<br>Patients with Impaired<br>Hepatic Function<br>[DHHS 2003] |
| Pregnancy test X | | X | | | | Х | Urine (or serum) pregnancy test (if WOCBP), as appropriate (see Protocol, Table 5) |

| | Screening<br>(up to | Check-<br>in | Trea | atment Pe<br>(Days) | riod | Follow-up<br>(10 [±5]<br>days | |
|---|---|---|---|---|---|---|---|
| Procedure <sup>1</sup> | 30 days<br>prior to<br>Day -1) | -1 | 1 | 1 2 | | postdose)<br>or Early<br>Termination | Notes |
| FSH | X | | | | | | Estradiol and FSH at<br>Screening (for women<br>of non-childbearing<br>potential), as<br>appropriate (see<br>Protocol, Table 5) |
| HIV antibody,<br>hepatitis B surface<br>antigen, and<br>hepatitis C antibody<br>testing | Х | | | | | If test has othe been performe 3 months befor drug administratesting at Screen not required | |
| Drug and alcohol screen | Х | Х | | | | | See Protocol, Table 5 |
| Laboratory<br>assessments<br>(include liver<br>chemistries) | Х | Х | | X | | X | Including serum<br>chemistry,<br>hematology, and<br>urinalysis. Results<br>from 24 hours after<br>dosing should be<br>available before<br>discharge on Day 3 |
| 12-lead ECG | Х | Х | Х | Х | Х | Х | See Section 10.1.2 for timing of assessments |
| Vital signs | Х | Х | X | Х | Х | Х | Respiratory rate and body temperature collected at Screening only See Section 10.1.2 for timing of assessments |
| Genetic sample | | Х | | | | | Informed consent for optional substudies (e.g., genetics research) must be obtained before collecting a PGx sample. The PGx sample can be collected anytime, but Day -1 is recommended |
| Study drug administration | | | Х | | | | |
| Blood collection for pharmacokinetics | | | Х | Х | Х | | See Section 10.1.2 for time points |

| | Screening (up to | Check-<br>in | Tre | atment Pe<br>(Days) | riod | Follow-up<br>(10 [±5] | Notes |
|---|---|---|---|---|---|---|---|
| Procedure <sup>1</sup> | 30 days<br>prior to<br>Day -1) | -1 | 1 | 2 | 3 | days postdose) or Early Termination | |
| Urine collection for pharmacokinetics | | | Х | Х | Х | | Participants with normal hepatic function and participants with hepatic impairment will have different collection intervals See Section 10.1.2 for time points |
| Saliva collection for pharmacokinetics | | | Χ | Х | Х | | See Section 10.1.2 for time points |
| AE/SAE review | Χ | Χ | <b>←========</b> | | X | | |
| Concomitant medication review | | Х | <b>←====</b> | | ·====> | Х | |

AE = adverse event, Clcr = estimated creatinine clearance; ECG = electrocardiogram, FDA = Food and Drug Administration; FSH = follicle-stimulating hormone; HIV = human immunodeficiency virus; PGx = pharmacogenetic, SAE = serious AE; WOCBP = women of childbearing potential.

When coinciding with safety and/or pharmacokinetic assessments, electrocardiograms, vital signs, and pharmacokinetic blood collections should be performed in said order.

#### 10.1.2. Protocol Defined Safety and PK Assessments

| Procedure <sup>1</sup> | | Treatment Period Time point (hours) | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Predose | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 6 | 8 | 12 | <b>24</b> <sup>2</sup> | 36 <sup>2</sup> | 48 <sup>2</sup> |
| 12-lead electrocardiogram | Х | | | | Х | Х | | | Х | | Х | Х | Χ | Χ | Х |
| Vital signs | Х | | | | Х | Χ | | | Χ | | Х | Χ | Χ | Χ | Χ |
| Study drug administration | | Χ | | | | | | | | | | | | | |
| Blood collection for pharmacokinetics | Х | | Х | Х | Χ | Х | Χ | Χ | Х | Х | Х | Х | Χ | Χ | Χ |
| Urine collection<br>for<br>pharmacokinetics<br>(participants with<br>normal hepatic<br>function) <sup>3</sup> | X | | | Х | | | Х | | х | Х | X | Х | Х | Х | Х |
| Urine collection<br>for<br>pharmacokinetics<br>(participants with<br>hepatic<br>impairment) <sup>4</sup> | X | | | | | X | | | | > | ( | x | x | х | х |
| Saliva collection | Χ | | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ |

When coinciding with safety and/or pharmacokinetic assessments, electrocardiograms, vital signs, and pharmacokinetic blood collections should be performed in said order.

The 24-, 36-, and 48-hour postdose time points correspond to time points on Day 2 and 3, respectively.

Urine collection intervals for participants with normal hepatic function (Group D and Group E, if applicable) include 0 (pre-dose), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours.

<sup>&</sup>lt;sup>4</sup> Urine collection intervals for participants with hepatic impairment (Group A, Group B, and Group C) include 0 hour (pre-dose), 0 to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 36, and 36 to 48 hours.

# 10.2. Appendix 2: Study Phases and Treatment Emergent Adverse Events

# 10.2.1. Study Phases

For Groups A, B, C, D, and E, assessments and events will be classified according to time of occurrence relative to the date/time of the study treatment.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date/Time < Study Treatment Date/Time |
| On-Treatment | Study Treatment Date/Time ≤ Date/Time ≤ Study Treatment Date/Time + 2 Days |
| Post-Treatment | Date/Time > Study Treatment Date/Time + 2 Days |

#### 10.2.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before enrollment date |
| Concomitant | Any medication that is not a prior |

#### NOTES:

• Please refer to Appendix 5: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

#### 10.2.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | If AE onset date/time is on or after treatment date/time & on or before the treatment stop date/time with 2 days lag time. |
| | <ul> <li>Study Treatment Date/Time ≤ AE Start Date/Time ≤ Study Treatment Date/Time</li> <li>+ 2 days.</li> </ul> |

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

#### 10.3.1. Reporting Process

#### Software

 SAS version 9.3 or higher and WinNonlin version software (version 9.3) and WinNonlin version 6.4 or higher will be used.

#### **Analysis Datasets**

- Analysis datasets will be created according CDISC standards SDTM IG Version 3.2 & ADaM IG Version 1.0.
- For creation of ADaM datasets (ADCM/ADCM1/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts described in the RAP.

#### 10.3.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the participant received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures (with the exception of individual PK
    concentration-time figures, where actual relative time will be used), summaries, statistical analyses
    and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures (mean figures only for PK concentrations), summaries and statistical analyses (excluding statistical analyses of PK parameters).

| Unscheduled Visits | |
|---|---|
| <ul> <li>Unscheduled visits will be considered when calculating baseline and in Table 2.9 and Table<br/>2.10, but will not be included in any other summary tables.</li> </ul> | |
| <ul> <li>Unscheduled visit</li> </ul> | Unscheduled visits will not be included in figures. |
| All unscheduled | All unscheduled visits will be included in listings. |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL State | Refer to IDSL Statistical Principals 7.01 to 7.13. |

# 10.3.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | centration Data |
|---|---|
| Descriptive Summary | Refer to IDSL PK Display Standards. |
| Statistics, Graphical | Refer to IDSL Statistical Principle 6.06.1. |
| Displays and Listings | For continuous data: |
| | <ul> <li>NQs at the beginning of a participant profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood.</li> <li>For NQs at the end of the participant profile (i.e. after the last incidence of a measurable concentration);</li> <li>for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can</li> </ul> |
| | erroneously indicate that absolutely no drug is present) |
| | <ul> <li>for summary statistics, these are set to 0 (to avoid skewing of the<br/>summary statistics)</li> </ul> |
| Pharmacokinetic Para<br>Descriptive Summary<br>Statistics, Graphical | Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly) If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual participant plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing). Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. Tameter Data N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CVb (%)) will be |
| Displays and Listings | reported. $CV_b$ (%) = $\sqrt{(exp(SD^2) - 1) * 100}$ |
| | (SD = SD of Ln-Transformed data) |
| Parameters Not<br>Being Ln-<br>Transformed | Tmax, tlag, CLr, lambda_z_lower, lambda_z_upper, and lambda_z_no. of points. |
| Parameters Not<br>Being Summarized | lambda_z_lower, lambda_z_upper, and lambda_z_no. of points. |
| Listings | Include the first point, last point and number of points used in the determination of |
| | λz and Rsq_adjusted for listings. |

#### 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from date of study drug administration (Dose Date):
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Dose Date → Study Day = Ref Date Dose Date</li>
  - Ref Data ≥ Dose Date → Study Day = Ref Date (Dose Date) + 1

#### 10.4.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Only the year of birth will be collected. The date and month will be imputed as PPD
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### 10.4.3. Safety

#### **ECG Parameters**

#### RR Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as:
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTeF} \right)^{3} \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **ECG Parameters**

• Machine read values of RR should not be replaced with derived values.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as:

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

# 10.5. Appendix 5: Reporting Standards for Missing Data

# 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including the follow-up visit.</li> <li>Withdrawn participants may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> <li>Early termination visits will be summarized as early termination visits.</li> </ul> |

10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

10.5.2.1. Handling of Missing and Partial Dates

| 10.5.2.1. | Hallulling of Missing and Partial Dates |
|---|---|
| Element | Reporting Detail |
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the date of study treatment; in this case the study treatment date will be used and hence the event is considered Treatment Emergent as per Appendix 2: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is more than 2 days after the date of study treatment; in this case the study treatment date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.6. Appendix 6: Values of Potential Clinical Importance

# 10.6.1. ECG

| ECG Parameter | Units | Potential Clinicall | Potential Clinically Important Range |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| | | > 450[1] | |
| Absolute QTc Interval | maga | > 450[2] | ≤ 479 <sup>[2]</sup> |
| ADSOIDLE QTC IIILEIVAI | msec | ≥ 480 <sup>[2]</sup> | ≤ 499[2] |
| | | ≥ 500 <sup>[2]</sup> | |
| Absolute PR Interval | msec | < 110 <sup>[1]</sup> | > 220[1] |
| Absolute QRS Interval | msec | < 75 <sup>[1]</sup> | > 110 <sup>[1]</sup> |
| Change from Baseline | | | |
| | msec | ≤ 30[2] | |
| Increase from Baseline QTc | msec | > 30[1] | ≤ 59 <sup>[2]</sup> |
| | msec | ≥ 60 <sup>[2]</sup> | |

#### NOTES:

- 1. Represent standard ECG values of PCI for HV studies.
- 2. Represent further subdivisions of ECG values for analysis.

# 10.6.2. Vital Signs

| Vital Sign Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.7. Appendix 7: Abbreviations & Trade Marks

# 10.7.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| Ae(t1-t2) | Amount of drug excreted in urine in a time intervals |
| Ae total | Total unchanged drug (total amount of drug excreted in urine) |
| AUC(0-∞) | Area under the concentration-time curve from time 0 (predose) extrapolated to infinite time |
| AUC(0-t) | Area under the concentration-time curve from time 0 (predose) to time of last quantifiable concentration |
| AUC(0-12) | Partial area under the curve estimated from urine concentrations samples collected from predose to 12 hours post dose |
| AUC(0-24) | Partial area under the curve estimated from urine concentrations samples collected from predose to 24 hours post dose |
| AUC(0-48) | Partial area under the curve estimated from urine concentrations samples collected from predose to 48 hours post dose |
| BMI | Body mass index |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL/F | Apparent oral clearance |
| CLr | Renal clearance of drug |
| Cmax | Maximum observed concentration |
| CVb | Coefficient of Variation (Between subjects) |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |
| fe% | Percentage of the given dose of drug excreted in urine |
| FDA | Food and Drug Administration |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| PCI | Potential Clinical Importance |
| PK | Pharmacokinetic(s) |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAUC(0-t) | The ratio of the AUC(0-t) observed in saliva relative to the AUC(0-t) in plasma |
| RAUC(0-∞) | The ratio of the AUC( $0-\infty$ ) observed in saliva relative to the AUC( $0-\infty$ ) in plasma |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| t1/2 | Terminal phase half life |
| | <u> </u> |

| Abbreviation | Description |
|---|---|
| λz | Terminal-phase rate constant |
| TFL | Tables, Figures & Listings |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| Tmax | Time to first occurrence of Cmax |
| Vz/F | Apparent volume of distribution of the terminal phase |

# 10.7.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

# 10.8. Appendix 8: List of Data Displays

# 10.8.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.10 | NA |
| Safety | 2.1 to 2.12 | NA |
| Pharmacokinetic | 3.1 to 3.11 | 3.1 to 3.11 |
| Section | Listi | ings |
| ICH Listings | 1 to | 40 |
| Other Listings | 41 to 46 | |

# 10.8.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.8.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| IA | Interim Analysis (Part 1) |
| SAC | Final Statistical Analysis Complete |

# 10.8.4. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition a | nd Populations | | | |
| 1.1. | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | SAC |
| 1.2. | Safety | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failures | | SAC |
| 1.4. | Screened | DV1 | Summary of Important Protocol Deviations | | SAC |
| Demog | raphics | | | | |
| 1.5. | Safety | DM1 | Summary of Demographic Characteristics | | SAC |
| 1.6. | Safety | DM5 | Summary of Race and Racial Combinations | | SAC |
| 1.7. | Safety | DM6 | Summary of Race and Racial Combinations Details | | SAC |
| 1.8. | Safety | DM11 | Summary of Age Ranges | | SAC |
| 1.9. | Safety | POP_T1 | Summary of Child-Pugh Scores | | SAC |
| Medica | Medical Conditions and Concomitant Medications | | | | |
| 1.10. | Safety | MH4 | Summary of Current Liver Disease and Cardiovascular Related Medical Conditions | | SAC |

# 10.8.5. Safety Tables

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events | | | | |
| 2.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | | SAC |
| 2.2. | Safety | AE1 | Summary of Drug-Related Adverse Events | | SAC |
| 2.3. | Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| 2.4. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| Labora | tory Values | | | | |
| 2.5. | Safety | LB1 | Summary of Clinical Chemistry Values Change from Baseline | | SAC |
| 2.6. | Safety | LB1 | Summary of Hematology Values Change from Baseline | | SAC |
| 2.7. | Safety | UR3 | Summary of Urinalysis Dipstick Results | | SAC |
| Electro | cardiograms | | | | |
| 2.8. | Safety | EG1 | Summary of ECG Findings | | SAC |
| 2.9. | Safety | SAFE_T1 | Summary of Frequency of Maximum Post-Dose ECG Parameter Corrected QTc Interval | | SAC |
| 2.10. | Safety | SAFE_T2 | Summary of Frequency of Maximum Change from Baseline for ECG Parameter Corrected QTc Interval | | SAC |
| 2.11. | Safety | EG2 | Summary of Change from Baseline in ECG Values | | SAC |
| Vital Si | gns | | | , | • |
| 2.12. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | SAC |

## 10.8.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| PK Cor | PK Concentration Data | | | | |
| 3.1 | PK Concentration | PKCT1 | Summary of Gepotidacin Plasma Pharmacokinetic<br>Concentration-Time Data (units) by Hepatic Function Group | | IA, SAC |
| 3.2 | PK Concentration | PKCT1 | Summary of Gepotidacin Urine Pharmacokinetic<br>Concentration-Time Data (units) by Hepatic Function Group | | IA, SAC |
| 3.3 | PK Concentration | PKCT1 | Summary of Gepotidacin Saliva Pharmacokinetic<br>Concentration-Time Data (units) by Hepatic Function Group | | IA, SAC |
| PK Par | ameters Tables | | | | |
| 3.4 | PK Parameter | PKPT4 | Summary of Derived Gepotidacin Plasma Pharmacokinetic Parameters by Hepatic Function Group | Parameters with units. If Group E are enrolled in part 2, then include a page of part 1 (Group B and D) alone in SAC deliverable as a reference for part 1 IA. | IA, SAC |
| 3.5 | PK Parameter | PKPT4 | Summary of Derived Gepotidacin Urine Pharmacokinetic Parameters by Hepatic Function Group | Parameters with units. | IA, SAC |
| 3.6 | PK Parameter | PKPT4 | Summary of Derived Gepotidacin Saliva Pharmacokinetic Parameters by Hepatic Function Group | Parameters with units. | IA, SAC |

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| PK Ana | llysis Tables | | | | |
| 3.7 | PK Parameter | РКРТ3 | Statistical Analysis of Gepotidacin Plasma Pharmacokinetic Parameters: Analysis of Variance (ANOVA) | AUC(0-∞) and Cmax only by Hepatic Function Group. If Group E are enrolled in part 2, then include a page of part 1 (Group B and D) alone in SAC deliverable as a reference for part 1 IA. | IA, SAC |
| 3.8 | PK Parameter | PKPT3 | Statistical Analysis of Gepotidacin Urine Pharmacokinetic Parameters: Analysis of Variance (ANOVA) | AUC(0-48) and CLr only by Hepatic Function Group. | IA, SAC |
| 3.9 | PK Parameter | PKPT3 | Statistical Analysis of Gepotidacin Saliva Pharmacokinetic Parameters: Analysis of Variance (ANOVA) | AUC(0-∞) and Cmax only by<br>Hepatic Function Group. | IA, SAC |
| 3.10 | PK Parameter | PK T1 | Statistical Analysis of Gepotidacin Plasma Tmax | | IA, SAC |
| 3.11 | PK Parameter | PK T1 | Statistical Analysis of Gepotidacin Saliva Tmax | | IA, SAC |

# 10.8.7. Pharmacokinetic Figures

| Pharmacokinetic : Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Concer | tration Plots | | | | |
| 3.1 | PK Concentration | PKCF1P | Individual Gepotidacin Plasma Concentration-Time Plots by Hepatic Function Group (Linear and Semi-Logarithmic) | Dashed line represents the LLQ. Present all hepatic function groups in the same plots. | IA, SAC |
| 3.2 | PK Concentration | PKCF1P | Individual Gepotidacin Urine Concentration-Time Plots by Hepatic Function Group (Linear and Semi- Logarithmic) | Dashed line represents the LLQ. Present all hepatic function groups in the same plots. Plot concentration at the collection midpoint. | IA, SAC |
| 3.3 | PK Concentration | PKCF1P | Individual Gepotidacin Saliva Concentration-Time Plots by Hepatic Function Group (Linear and Semi- Logarithmic) | Dashed line represents the LLQ. Present all hepatic function groups in the same plots. | IA, SAC |
| 3.4 | PK Concentration | PKCF2 | Mean Gepotidacin Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | Dashed line represents the LLQ. Present all treatment groups in the same plots. | IA, SAC |
| 3.5 | PK Concentration | PKCF2 | Mean Gepotidacin Urine Concentration-Time Plots (Linear and Semi-Logarithmic) | Dashed line represents the LLQ. Present all treatment groups in the same plots. Plot concentration at the collection midpoint. | IA, SAC |
| 3.6 | PK Concentration | PKCF2 | Mean Gepotidacin Saliva Concentration-Time Plots (Linear and Semi-Logarithmic) | Dashed line represents the LLQ. Present all treatment groups in the same plots. | IA, SAC |

| Pharma | cokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.7 | PK Concentration | PKCF3 | Median Gepotidacin Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) | Dashed line represents the LLQ. Present all treatment groups in the same plots. | IA, SAC |
| 3.8 | PK Concentration | PKCF3 | Median Gepotidacin Urine Concentration-Time Plots (Linear and Semi-Logarithmic) | Dashed line represents the LLQ. Present all treatment groups in the same plots. Plot concentration at the collection midpoint. | IA, SAC |
| 3.9 | PK Concentration | PKCF3 | Median Gepotidacin Saliva Concentration-Time Plots (Linear and Semi-Logarithmic) | Dashed line represents the LLQ. Present all treatment groups in the same plots. | IA, SAC |
| Explora | tory Objectives | 1 | | | |
| 3.10 | PK Concentration | PK_F4 | Scatter Plot of Gepotidacin Saliva and Unbound Plasma<br>Concentrations by Hepatic Function Group | Present all treatment groups in the same plots. | IA, SAC |
| 3.11 | PK Parameter | PK_F5 | Scatter Plot of Gepotidacin Saliva and Unbound Plasma PK Parameters by Hepatic Function Group | Present all treatment groups in the same plots. Repeat for PK parameters AUC(0-t), AUC(0-inf), Cmax, CL/F and t½. | IA, SAC |
| 3.12 | PK Concentration | PK_F4 | Scatter Plot of Gepotidacin Saliva and Total Plasma<br>Concentrations by Hepatic Function Group | Present all treatment groups in the same plots. | IA, SAC |
| 3.13 | PK Parameter | PK_F5 | Scatter Plot of Gepotidacin Saliva and Total Plasma PK Parameters by Hepatic Function Group | Present all treatment groups in the same plots. Repeat for PK parameters AUC(0-t), AUC(0-inf), Cmax, CL/F and t½. | IA, SAC |

# 10.8.8. ICH Listings

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Group | Assignment | | | | · |
| 1. | Safety | TA1 | Listing of Planned and Actual Group | | SAC |
| Subjec | t Disposition | | | | |
| 2. | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC |
| 3. | Screened | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 4. | Screened | DV2 | Listing of Important Protocol Deviations | | SAC |
| 5. | Safety | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| 6. | Enrolled | SP3 | Listing of Subjects Excluded from Any Population | | SAC |
| 7. | Safety | SAFE_L1 | Listing of Subjects in Previous Clinical Trial | | SAC |
| Demog | raphics and Ba | seline Characteri | stics | | |
| 8. | Safety | DM4 | Listing of Demographic Characteristics | | SAC |
| 9. | Safety | DM10 | Listing of Race | | SAC |
| 10. | Safety | SAFE_L2 | Listing of Child-Pugh Scores | | SAC |
| Concor | mitant Medicati | ons | | | · |
| 11. | Safety | MH2 | Listing of Cardiovascular and Liver Disease Related Medical Conditions | | SAC |
| 12. | Safety | CM3 | Listing of Concomitant Medications | | SAC |
| Exposu | ure | | | | |
| 13. | Safety | SAFE_L3 | Listing of Exposure Data | | SAC |

| ICH : L | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events | | | | · |
| 14. | Safety | AE2 | Listing of Relationship Between System Organ Class and Verbatim Text | | SAC |
| 15. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 16. | Safety | AE8 | Listing of All Adverse Events | | SAC |
| 17. | Safety | AE8 | Listing of Study Drug Related Adverse Events | | SAC |
| 18. | Safety | SAFE_L4 | Listing of Serious Adverse Events (Fatal and Non-Fatal) | | SAC |
| 19. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study | | SAC |
| 20. | Safety | SAFE_L5 | Listing of Liver Adverse Events | Conditional Display | SAC |
| 21. | Safety | SAFE_L6 | Listing of Cardiovascular Adverse Events | Conditional Display | SAC |
| Labora | tory Values | | | | |
| 22. | Safety | SAFE_L7 | Listing of Clostridium Difficile Testing | | SAC |
| 23. | Safety | LB5 | Listing of Clinical Chemistry Toxicities of Grade 3 or Higher | | SAC |
| 24. | Safety | LB5 | Listing of All Clinical Chemistry Data for Subjects with Toxicities of Grade 3 or Higher | | SAC |
| 25. | Safety | LB5 | Listing of Hematology Toxicities of Grade 3 or Higher | | SAC |
| 26. | Safety | LB5 | Listing of All Hematology Data for Subjects with Toxicities of Grade 3 or Higher | | SAC |
| 27. | Safety | UR2a | Listing of Urinalysis Toxicities of Grade 3 or Higher | | SAC |
| 28. | Safety | UR2a | Listing of All Urinalysis Data for Subjects with Toxicities of Grade 3 or Higher | | SAC |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Electrocardiograms | | | | | |
| 29. | Safety | EG5 | Listing of Abnormal ECG Findings | | SAC |
| 30. | Safety | EG5 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | SAC |
| 31. | Safety | EG3 | Listing of ECG Values of Potential Clinical Importance | | SAC |
| 32. | Safety | EG3 | Listing of All ECG Values for Subjects with any Value of Potential Clinical Importance | | SAC |
| Vital Si | Vital Signs | | | | |
| 33. | Safety | VS4 | Listing of Vital Signs of Potential Clinical Importance | | SAC |
| 34. | Safety | VS4 | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | | SAC |
| Liver E | vent | | | | <u>'</u> |
| 35. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | Conditional Display | SAC |
| 36. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping<br>Events | Conditional Display | SAC |
| 37. | Safety | SAFE_L8 | Listing of Alcohol Intake at Onset of Liver Event | Conditional Display | SAC |
| 38. | Safety | PKCL1X | Listing of Plasma Concentration Data for Subjects with Liver Stopping Events | Conditional Display | SAC |
| 39. | Safety | LIVER7 | Listing of Liver Biopsy Details | Conditional Display | SAC |
| 40. | Safety | LIVER8 | Listing of Liver Imaging Details | Conditional Display | SAC |

# 10.8.9. Non-ICH Listings

| Other (non-ICH): Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Pharmacokinetic | | | | | |
| 41. | PK<br>Concentration | PKCL1P | Listing of Plasma Gepotidacin Concentrations (units) by Hepatic Function Group | Please list all the concentration data including unscheduled. Repeat for all Hepatic Function Groups. | IA, SAC |
| 42. | PK<br>Concentration | PKUL1P | Urine Gepotidacin Concentrations by Hepatic Function | Please list all the concentration data including unscheduled. Repeat for all Hepatic Function Groups. | IA, SAC |
| 43. | PK<br>Concentration | PKCL1X | Saliva Gepotidacin Concentrations by Hepatic Function | Please list all the concentration data including unscheduled. Repeat for all Hepatic Function Groups. | IA, SAC |
| 44. | PK Parameter | PKPL1P | Listing of Gepotidacin Plasma Pharmacokinetic Parameters by Treatment | | IA, SAC |
| 45. | PK Parameter | PKPL1P | Listing of Gepotidacin Urine Pharmacokinetic Parameters by Treatment | | IA, SAC |
| 46. | PK Parameter | PKPL1P | Listing of Gepotidacin Saliva Pharmacokinetic Parameters by Treatment | | IA, SAC |